CLINICAL TRIAL: NCT04946500
Title: Clindamycin in Prosthetic Joint Infections Caused by Staphylococcus
Brief Title: Clindamycin in Prosthetic Joint Infections Caused by Staphylococcus (CISTA)
Acronym: CISTA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CISTA - 29BRC21.0123
Record Dates: First submitted 2021-05-06; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-04

CONDITIONS: Prosthetic Joint Infection; Staphylococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clindamycin and Rifampicin: Patients treated with Clindamycin and Rifampicin
- Clindamycin and Fluoroquinolone: Patients treated with Clindamycin and Fluoroquinolone

SUMMARY:
The alternatives to the combination of Fluoroquinolone and Rifampicin in prosthetic joint infections (PJI) caused by staphylococcus are currently unclear. Clindamycin is prescribed as dual therapy in this indication, and provides many advantages. We conducted a multicenter retrospective observational study evaluating the efficacy and safety of Clindamycin in prosthetic joint infections due to staphylococcus between January 2013 and December 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PJI defined according to the IDSA.
* Infection must be mono-microbial or multi-microbial with Staphylococcus spp sensitive to Clindamycin.
* Infection may be acute or chronic, nosocomial or community-acquired.
* Patient having received a curative treatment with Clindamycin.

Exclusion Criteria:

* Patients with osteitis, osteomyelitis, septic arthritis in native joints, diabetic foot infections, spondylodiscitis, infections in external fixator, surgical site infections following neurosurgical management, bedsores, skin and soft tissue infections.
* Patients with mono-microbial infections other than Staphylococcus, multi-microbial infections including other bacteria than Staphylococcus, suspected Osteoarticular Infection without microbial identification.
* Patients with clindamycin-resistant Staphylococcal PJI, constitutive MLSb phenotype.
* Patients having received suspensive treatment with Clindamycin.
* Patients treated with Clindamycin as last line of treatment for a duration of less than 14 days.
* Patients refusing to participate
* Patients under legal protection (guardianship, curatorship, ..)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Prosthetic Joint Infections caused by Staphylococccus treated with Clindamycin
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Failure of Clindamycine | within 2 years of the diagnosis (within one year for patients diagnosed in December 2019)
  New diagnosis of PJI at the same site, caused by the same microbial agent

SECONDARY OUTCOMES:
Safety of Clindamycin | During the treatment and 6 month after
  Safety of Clindamycin in the treatment of PJI
Correlation between failure of Clindamycin and blood level of Clindamycin | within 2 years of the diagnosis (within one year for patients diagnosed in December 2019)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three month and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.